CLINICAL TRIAL: NCT04901910
Title: Social Media Intervention for Cannabis Use and Physical Activity in Emerging Adults - Physical Activity
Brief Title: Social Media Intervention - Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Erin Bonar, Associate Professor of Psychiatry, Medical School and Adjunct Associate Professor of Psychology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00195927
Record Dates: First submitted 2021-05-14; First posted 2021-05-26 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Cannabis Use
Keywords: social media
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Physical Activity (PA) Social Media Group (Experimental): This will be an 8 week Social Media Group available to the participant focused on health and well-being.
  Interventions: Behavioral: Physical Activity (PA) Social Media Group
- Verdi plus PA Social Media Group (Experimental): This will be an 8 week Social Media Group available to the participant focused on health and well-being.
  Interventions: Behavioral: Verdi plus PA Social Media Group
- Attention-Control condition Social Media Group (No Intervention): This will be an 8 week Social Media Group available to the participant with social media topics.

INTERVENTIONS:
Behavioral: Physical Activity (PA) Social Media Group — Participants will have access to the secret Social Media page that will deliver health information focused on increasing healthy activities and well-being. This information will be posted by e-coaches. Participants can interact with the e-coaches as well as other study members in the group.
  Arms: Physical Activity (PA) Social Media Group
Behavioral: Verdi plus PA Social Media Group — Participants will have access to the secret Social Media page that will deliver health information focused on increasing healthy activities, well-being, and reducing risky behaviors. This information will be posted by e-coaches. Participants can interact with the e-coaches as well as other study members in the group.
  Arms: Verdi plus PA Social Media Group

SUMMARY:
The purpose of the study is to develop and test social media interventions to help young people increase well-being and reduce risky behaviors. The study will help us learn about ways to deliver wellness information in a way that is appealing and helpful to young people that use social media.

Eligible participants will be enrolled after baseline survey is completed. Participants will be involved with the secret social media group they are assigned to for 8 weeks. In addition, surveys will be completed at various times during and after the 8 week social media group.

ELIGIBILITY:
Inclusion Criteria:

* self-report using cannabis at least 3 times per week or more often in the past month
* active Facebook profile

Exclusion Criteria:

* participants who cannot read English will be informally excluded
* if participants fail identity verification based on:

  * Internet Protocol (IP) addresses
  * survey time completion
  * repeat attempts
  * survey responses
  * photo identification from a time stamped self picture sent to the research team
* cannot safely engage in moderate to vigorous physical activity [assessed at screening]
* participated in previous Project Verdi waves

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-05-18 (Actual); Primary Completion 2021-12-25 (Actual); Study Completion 2021-12-25 (Actual)

PRIMARY OUTCOMES:
Acceptability of intervention (i.e., ratings of e-coaches, ) | 3 months (after baseline)
  Acceptability ratings completed by participants:
  How helpful were the e-coaches?
  1. Not at all
  2. A little
  3. Somewhat
  4. Very Much
  5. Extremely
Acceptability of intervention (i.e., helpfulness of peer interaction) | 3 months (after baseline)
  Acceptability ratings completed by participants:
  How helpful was it to interact with other peers in the group?
  1. Not at all
  2. A little
  3. Somewhat
  4. Very Much
  5. Extremely
Feasibility of intervention as evidenced by metrics of key activities (accepting group invitation) | 8 weeks post-group start
  number/percent who accept group invite
Feasibility of intervention as evidenced by metrics of key activities (engaging in the group) | 8 weeks post-group start
  number/percent who comment engage (i.e., comment at least one time)

CONTACTS AND LOCATIONS:
Overall Officials: Erina Bonar, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bonar EE, Chapman L, Pagoto S, Tan CY, Duval ER, McAfee J, Collins RL, Walton MA. Social media interventions addressing physical activity among emerging adults who use cannabis: A pilot trial of feasibility and acceptability. Drug Alcohol Depend. 2023 Jan 1;242:109693. doi: 10.1016/j.drugalcdep.2022.109693. Epub 2022 Nov 11. PMID 36442441